CLINICAL TRIAL: NCT03290820
Title: Aspirin Improve Survival of Patients With N2-3 Nasopharyngeal Carcinoma: A Phase 2 Prospective Randomized Controlled Trial
Brief Title: Aspirin Improve Survival of N2-3 Nasopharyngeal Carcinoma Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yun-fei Xia, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-FXY-067
Record Dates: First submitted 2017-09-13; First posted 2017-09-25 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; N2-3 disease; distant metastasis; aspirin; survival
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy; Aspirin

STUDY DESIGN:
Intervention Model Description: The patients eligible are divided randomly. All the patients will receive concurrent chemoradiotherapy. The cases in the Experimental Group will receive daily aspirin of 75mg.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controlled Group (Active Comparator): The patients in the Controlled Group are allocated to receive radiotherapy and concurrent chemotherapy.
  Interventions: Radiation: Radiotherapy; Drug: Concurrent chemotherapy
- Experimental Group (Experimental): The patients in the Experimental Group are allocated to receive radiotherapy and concurrent chemotherapy plus daily aspirin.
  Interventions: Radiation: Radiotherapy; Drug: Concurrent chemotherapy; Drug: Aspirin

INTERVENTIONS:
Radiation: Radiotherapy — Technique: intensity-modulated radiotherapy; Dose: GTVnx 6810cGy/30Fr, GTVnd 6400-6600cGy/30Fr, CTV1 6000cGy, CTV2 5400cGy.
Drug: Concurrent chemotherapy — Nedaplatin 80mg/m2 d1+5-flurouracil 500mg/m2 d2-5, every 3 weeks; a total of 2-3 cycles.
Drug: Aspirin — Daily aspirin of 75mg, from the starting date of radiotherapy.
  Arms: Experimental Group

SUMMARY:
Nasopharyngeal carcinoma (NPC) is one of the most common maligancies of China. In the era of intensity-modulated radiotherapy (IMRT), the 5-year overall survival (OS) has now reached 85.0% or more. However, even after chemoradiation, the 5-year distant-metastasis rate of patients with N2-3 NPC is still 36.7%. Aspirin is proven in lab and clinical studies to have the abilities of inhibiting the inflammation which could enhance metastasis of breast and colorectal cancers. And before this study, it was discovered that regular aspirin intake might be associated with distant-metastasis-free survival (MFS) and OS independently. So this Phase 2 trial was conducted to validate the impact of aspirin on prognosis of N2-3 NPC.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is one of the most common maligancies of China. In the era of intensity-modulated radiotherapy (IMRT), the 5-year overall survival (OS) has now reached 85.0% or more. However, the prognosis of the patients with late N (N2-3) diseases remains poor. Even after chemoradiation, the 5-year distant-metastasis rate of these patients is nearly 36.7%. Additionally, these patients occupies about 30.0% of the whole NPC population. To improve the prognosis of the patients with N2-3 NPC, there is a need to explore a new, practical and effective method to eliminate the distant metastasis.

Aspirin is proven in lab and clinical studies to have the abilities of inhibiting the inflammation which could enhance metastasis of many malignant tumors, such as breast and colorectal cancers. And before this study, patients with N2-3 nonmetastatic NPC between 2008 and 2011 were retrospectively analyzed, to discovered that regular aspirin intake might be associated with distant-metastasis-free survival (MFS) and OS independently. So this Phase 2 randomized controlled trial was conducted to validate the impact of aspirin on prognosis of N2-3 NPC.

This study aim to enroll patients with T1-4N2-3M0 NPC. All the patients will be treated with IMRT and concurrent chemotherapy of the PF (Nedaplatin + 5-flurouracil) regimen. After randomization, patients in the Experimental Group will also receive daily aspirin of 75mg. The 5-year MFS is the primary endpoint. And the 5-year OS and aspirin-related toxicities are the secondary endponits.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic dianosis of nasopharyngeal carcinoma
* Stage of T1-4N2-3M0 (UICC/AJCC classification ver. 7)
* 18-70 years old
* Karnofsky performance score > 70

Exclusion Criteria:

* Distant metastasis before or during radiotherapy
* Severe dysfunctions of liver, kidney, lung, heart of bone marrow which are not fit for radiotherapy
* Prior malignancies
* Prior history of radiotherapy, chemotherapy or monoclonal antibody therapy
* Participation of other drug trials within 3 months
* Regular use of aspirin before dianosis
* Contraindication or allergy of aspirin
* Patients who are considered by the researchers not suitable to participate this trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Distant-metastasis-free survival | 5 years after diagnosis
  The percentage of patients of a data set who survive without distant metastasis after a defined period of time from pathologic diagnosis

SECONDARY OUTCOMES:
Overall survival | 5 years after diagnosis
  The percentage of patients of a data set who survive after a defined period of time from pathologic diagnosis
Aspirin-related toxicities | 5 years after diagnosis
  Incidence of aspirin-related toxicities such as gastrointestinal bleeding and liver dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Yun-fei Xia, M.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No